CLINICAL TRIAL: NCT02793960
Title: A Phase 1 Study to Evaluate the Safety, Pharmacokinetics and Therapeutic Effect of Topical BPM31510 3.0% Cream in Patients With Epidermolysis Bullosa
Brief Title: Topical BPM31510 3.0% Cream in Patients With Epidermolysis Bullosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shasa Hu (Other)
Collaborators: BPGbio (Industry)
Responsible Party: Sponsor-Investigator, Shasa Hu, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20151103
Record Dates: First submitted 2016-05-18; First posted 2016-06-08 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical BPM31510 3.0% Cream (Experimental): Patients/ caregiver will apply topical BPM31510 3.0% cream from every other day to twice per week to wounded skin, and every day to a section of intact skin for up to 12 weeks.The area to be covered may not exceed 10% BSA inclusive of intact skin area, and other lesions.
  Interventions: Drug: topical BPM31510 3.0% Cream

INTERVENTIONS:
Drug: topical BPM31510 3.0% Cream — Application of drug to lesions of epidermolysis bullosa

SUMMARY:
This is a single-center study to investigate the effects of a topical cream on patients 12 years of age and older that have been diagnosed with epidermolysis bullosa.

DETAILED DESCRIPTION:
The trial will be conducted in patients with any form of Epidermolysis Bullosa (EB) with at least 1 active EB wound between 2.5 and 50 cm2 in size or up to 10% of the Body Surface Area. The investigators will identify an "index lesion" and other lesions for treatment An area of un-involved skin will also be treated with the study cream. This are will be used for testing by producing tiny blisters th so that the underlying tissue can be examined using a special microscope.

Patients will apply the study cream

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 12 years of age at the time of screening.
2. Have primary, histologically confirmed EB verified by immunofluorescent antigenic mapping (EM) prior to starting application of study drug
3. Have no other dermatological disease that may adversely impact wound healing.
4. Willing to refrain from using topical creams or lotions other than the study drug to the designated areas during the treatment period and from washing the designated areas until the next application is done.
5. Willing to refrain from exposure to excessive direct sunlight or ultraviolet light for the duration of the study.
6. Laboratory values for the tests listed in the Study Schedule are within the local reference ranges as defined by the local laboratory, or "out of range" test results are clinically acceptable to the investigator. Acceptable "out of range" values are generally those within the patient's normal baseline levels due to concurrent medications or disease processes with the exception of INR and PT/APTT.
7. Caregiver/guardian or patient is able to follow study required instructions and likely to complete all study visit requirements.
8. Has a provided written informed consent by patient or a legal guardian, including consent for tissue to be examined and stored by the Department of Dermatology and Cutaneous Surgery. If the patient is between 12 and 17 years of age, assent must be given by the patient.
9. Guardian has provided written consent to allow photographs of the target EB lesion(s) to be used as part of the study data and documentation.
10. Females of childbearing potential must have a negative urine or serum pregnancy test at screening and be using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy).
11. Have an INR value of 0.8-1.2 as well as normal PT/APTT.
12. With at least 1 active EB wound between 2.5 and 50 cm2 in size on nonflexual surfaces

Exclusion Criteria:

1. Received systemic therapy of living skin equivalent grafting in the past 30 days prior to baseline visit.
2. Known or suspected systemic cancer such as lymphoma or leukemia.
3. Evidence of dermatological disease or confounding skin condition in the treatment area, e.g., BCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, xerodermapigmentosa, or clinical evidence of infection.
4. Concurrent disease or treatment that suppresses the immune system.
5. Any chronic medical condition that, in the judgment of the investigator(s), can interfere with the performance of the study or would place the patient at undue risk.
6. Known sensitivity to any of the ingredients in the trial medication (BPM31510 3.0% Cream
7. Treatment with any systemic immunomodulators or immunosuppressants within the 2 months prior to enrollment, for a duration longer than 2 weeks.
8. Use of any topical immunomodulators such as topical tacrolimus.
9. Use of systemic or topical steroids within 30 days prior to enrollment is excluded (inhaled steroids and ophthalmic drops containing steroids are allowed).
10. Any elective or non-elective surgery other than biopsy for EB, or surgeries for the treatment of sequelae of EB such as g-tube placement or esophageal dilatation within 4 weeks prior to enrollment during the study. Elective procedures pertaining to skin graft will not be allowed at any time.
11. Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of enrollment.
12. In the investigator's opinion, evidence of unwillingness or inability of the patient or caregiver to follow the restrictions and complete the study.
13. Has any clotting disorder, or is being treated with any anticoagulant.
14. Any abnormal laboratory value or concurrent illness that, in the opinion of the investigator, should preclude the patient's participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 16 weeks
  Analysis of laboratory values and/or Adverse events

SECONDARY OUTCOMES:
Peak Plasma Concentration of BPM31510 | Day 1, Day 3, week 8.
  Blood will be drawn pre-study drug application on Day 1 and post study drug application on Day 3 and Week 8
Decrease in VAS Pain Scale questionnaire | Baseline, 16 weeks
  Subject completed Questionnaire will assess the .pain at each visit.
Change in Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) | Baseline, 16 weeks
  The (EBDASI) be utilized by investigators to quantify wound healing and scarring at each visit.
Change in the Lansky Performance Scale and the Children's Dermatology Life Quality Index | Baseline, 16 weeks
  Subject completed questionnaires will be completed at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Department of Dermatology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No